CLINICAL TRIAL: NCT02869321
Title: Evaluation of Analgesic Efficacy of Transmucosal Fentanyl for Breakthrough Pain Caused by Interventional Gastrostomy
Brief Title: Analgesic Efficacy of Transmucosal Fentanyl for Breakthrough Pain Caused by Interventional Gastrostomy
Acronym: ANTALGIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2014-003352-32
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2018-05

CONDITIONS: Gastrostomy; Breakthrough Pain; Upper Aerodigestive Tract Neoplasms
MeSH Terms: conditions — Breakthrough Pain; Head and Neck Neoplasms | interventions — Fentanyl; Morphine; Gastrostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): Administration of Morphine Sulfate Placebo and Fentanyl
  1. Morphine Sulfate Placebo: oral solution administered through nasogastric tube, 10% of daily dose of morphine of background treatment, 1 hour before gastrostomy
     +
  2. Fentanyl: nasal spray solution, 100 µg pulverisation, 15 min before gastrostomy, if not efficacy second dose after 15 min during gastrostomy
  Administration 1+2 if pain after 4 hours from gastrostomy
  Interventions: Drug: Fentanyl; Drug: Morphine Sulfate placebo; Procedure: Gastrostomy
- Morphine Sulfate (Placebo Comparator): Administration of Morphine Sulfate and Fentanyl Placebo
  1. Morphine Sulfate: oral solution administered through nasogastric tube, 10% of daily dose of morphine of background treatment, 1 hour before gastrostomy
     +
  2. Fentanyl Placebo: nasal spray solution, 100 µg pulverisation, 15 min before gastrostomy, if not efficacy second dose after 15 min during gastrostomy
  Administration 1+2 if pain after 4 hours from gastrostomy
  Interventions: Drug: Morphine Sulfate; Drug: Fentanyl placebo; Procedure: Gastrostomy

INTERVENTIONS:
Drug: Fentanyl
  Other Names: PECFENT®
  Arms: Fentanyl
Drug: Morphine Sulfate
  Other Names: ORAMORPH®
  Arms: Morphine Sulfate
Drug: Fentanyl placebo
  Arms: Morphine Sulfate
Drug: Morphine Sulfate placebo
  Arms: Fentanyl
Procedure: Gastrostomy

SUMMARY:
Patients with Head & Neck Squamous Cell Carcinoma often need a gastrostomy. It can be performed with a radiological approach. This procedure is usually not performed under general anesthesia, but local anesthesia is not sufficient to counteract pain due to gastric insufflation and incision of the abdominal wall. Standard analgesic treatments are usually not well-fitted due to onset of action or route of administration. An alternative solution could be fentanyl nasal spray, a treatment with a fast onset of action and with easy use allowing repetition if needed, during the procedure.

The purpose of this study is to compare analgesic efficacy of nasal instillation of PECFENT® to usually administered morphinic analgesic treatment with fast onset of action (ORAMORPH®), in radiologic percutaneous gastrostomy tube placement:

* during the procedure
* following the procedure (measured by Visual Analog Scale (VAS) for Pain at 15 min, 30 min, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 12 hours after procedure).

Secondary purposes are to compare easiness of 2 treatments and their adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient care for cancer of the upper aerodigestive tract (except sinonasal)
* > 18, all weights, all sexes
* Under balanced background opioid treatment since longer than 7 days (VAS < 5)
* Needing a radiologic gastrostomy under local anesthesia
* Informed consent
* Affiliation to social security plan
* Preliminary medical examination

Exclusion Criteria:

* Non balanced morphinic treatment : modification of analgesic treatment during 7 previous days
* Radiotherapy of nasal fossae/sinus
* Technical impossibility or contraindication to PECFENT®, ORAMORPH® and associated drugs
* Impossibility of pain evaluation by patient
* Belonging to protected class: pregnant or breastfeeding woman, person deprived of liberty for judiciary or administrative decision, under-18, person under legal protection or incapable of giving consent, person in life-and-death emergency incapable of giving a preliminary consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Intensity of breakthrough pain during the gastrostomy | during gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 15 min after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 30 min after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 1 hour after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 2 hours after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 3 hours after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 4 hours after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 6 hours after gastrostomy
  Pain measured by VAS
Intensity of pain following the gastrostomy | 12 hours after gastrostomy
  Pain measured by VAS
Necessity of a second analgesic treatment after gastrostomy | up to 12 hours from gastrostomy
  in case of Pain VAS >4

SECONDARY OUTCOMES:
Evaluation of satisfaction of patient with analgesic efficacy | up to 1 day from gastrostomy
  Questionnaire
Evaluation of satisfaction of staff with analgesic efficacy and easiness to use of treatments | up to 1 day from gastrostomy
  Questionnaire
Compliance of times of administration of treatments with the procedure | day 0
Comparison of adverse effects of administered drugs | up to 24 hours post gastrostomy

CONTACTS AND LOCATIONS:
Overall Officials: Patrice GALLET, Principal Investigator — Service ORL - CHU NANCY - France
Locations (1):
- Service ORL - CHU NANCY, Nancy, France

IPD SHARING:
Plan to Share IPD: No